CLINICAL TRIAL: NCT00844714
Title: Cardiovascular Risk Markers in Patients With Rheumatoid Arthritis: Effect of Rituximab Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RITUXANFMD
Record Dates: First submitted 2009-02-12; First posted 2009-02-16 (Estimated); Results first posted 2014-06-23 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-05

CONDITIONS: Endothelial Function; Rheumatoid Arthritis; Inflammation
Keywords: endothelial function; rheumatoid arthritis; cardiovascular risk; rituxan therapy
MeSH Terms: conditions — Arthritis, Rheumatoid; Inflammation | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituxan (Experimental)
  Interventions: Drug: Rituxan

INTERVENTIONS:
Drug: Rituxan — 1000mg rituxan by intravenous infusion will be given on day 1 and day 15 of the study

SUMMARY:
The purpose of this investigation is to determine the effects of Rituxan therapy in individuals with rheumatoid arthritis on endothelial function and other markers of endothelial function

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give written informed consent and comply with the requirements of the study protocol
* Negative serum pregnancy test (for women of child bearing age)
* Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for twelve months (1 year) after completion of treatment.
* IgG & IgM levels within normal limits
* Adequate renal function as indicated by serum creatinine measurements.
* No previous biological use (investigational or approved) except for the three approved anti-TNF alpha therapies
* Patients who have been treated with anti-TNF alpha therapies must be off of infliximab and adalimumab for two months before study entry and off of etanercept for one month before study entry
* No use of phosphodiesterase type 5 inhibitors (PDE5) (i.e. Sildenafil, Tadalafil, and Vardenafil) 1 week prior to the study and during the course of the study.
* SBP ≤ 140/90 for two months prior to study enrollment

Exclusion Criteria:

* Prior history of MI, CVA, CABG, PTCA, or peripheral vascular disease
* Any serious concomitant medical condition that could interfere with the study.
* Patients with insulin dependent diabetes
* Failure to provide written consent.
* Individuals with HIV infections
* SBP > 140/90 at two months prior to study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-11; Primary Completion 2012-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Hsue PY, Scherzer R, Grunfeld C, Imboden J, Wu Y, Del Puerto G, Nitta E, Shigenaga J, Schnell Heringer A, Ganz P, Graf J. Depletion of B-cells with rituximab improves endothelial function and reduces inflammation among individuals with rheumatoid arthritis. J Am Heart Assoc. 2014 Oct 21;3(5):e001267. doi: 10.1161/JAHA.114.001267. PMID 25336464

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituxan: Rituxan: 1000mg rituxan by intravenous infusion on day 1 and day 15
Period: Overall Study
Arm/Group | Rituxan
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: per protocol, patients with active rheumatoid arthritis (RA) who had high levels of systemic inflammation
Arm/Group | Rituxan
Number analyzed (Participants) | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54 [46 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 20
Flow-mediated vasodilation (FMD) [Median (Inter-Quartile Range); unit: mm] — endothelial function as assessed by flow-mediated vasodilation of the brachial artery
  mm | 3.9 [3.4 to 5.8]

OUTCOME MEASURES:

1. Primary Outcome: Flow-mediated Vasodilation (FMD)
Description: endothelial function as assessed by flow-mediated vasodilation of the brachial artery
Time Frame: 12 weeks, 24 weeks
Measure: Median (Inter-Quartile Range); unit: percentage change in diameter
Arm/Group | Rituxan
Number analyzed (Participants) | 20
percentage change in diameter
  12 weeks | 6.1 [4.9 to 7.6]
  24 weeks | 4.4 [3.3 to 6.1]

ADVERSE EVENTS:
Arm/Group | Rituxan
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes